CLINICAL TRIAL: NCT00427050
Title: An Open-label, Multi-centre, Dose-escalation, Cohort Study to Determine the Optimal Tolerated Regime and Safety of PEP005 Topical Gel When Applied to a 25 cm2 Contiguous Actinic Keratoses Treatment Area on the Face or Face and Scalp.
Brief Title: A Study to Determine the Optimal Tolerated Regime and Safety of PEP005 Topical Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-007
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2008-12

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses (AK); PEP005; Topical; Dermatology
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

INTERVENTIONS:
Drug: PEP005

SUMMARY:
The purpose of this study is to determine the optimal tolerated regime of PEP005 for the treatment of actinic keratoses of the face or face and scalp.

DETAILED DESCRIPTION:
Actinic keratoses (AK) is a common skin condition characterized by rough, scaly patches or sores on the top layer of the skin which if left untreated can progress to skin cancer. Current treatments can cause scarring and hypopigmentation, be inconvenient, or require long treatment duration. Non-invasive alternative therapy for treatment of AK lesions is thus being researched.

ELIGIBILITY:
1. Male patients at least 18 years of age.
2. Post-menopausal female patients i.e., no menses for at least 12 consecutive months, or without a uterus.
3. Four to eight clinically typical, visible and discrete AK lesions within a contiguous 25 cm2 treatment area on the face or face and scalp.

5. Ability to follow study instructions and likely to complete all study requirements.

6. Written informed consent has been obtained. 7. Agreement from the patient to allow photographs of the selected AK treatment area to be taken and used as part of the study data package.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Optimal tolerated regime of PEP005 Topical Gel in patients, when administered as either two day or three day application schedules to a 25 cm2 contiguous AK treatment area on the face or face and scalp

SECONDARY OUTCOMES:
Efficacy at 2 or 3day application PEP005 Topical Gel at the MTD of 0.025% in the Expanded Cohort, and at 2 lower concs of 0.0175% and 0.0125% at either a 2 or 3day application, when applied to 25cm2 AK treatment area on face or face/scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Katsamas, Study Director — Peplin Operations Pty Ltd
Locations (9):
- Australia (6):
  - Skin and Cancer Foundation, Darlinghurst, New South Wales
  - Southderm Pty Ltd, Kogarah, New South Wales
  - St George Dermatology and Skin Cancer Centre, Level 3, 22 Belgrave St, Kogarah, New South Wales
  - South East Dermatology, Belmont Specialist Centre, 1202 Creek Rd, Carina Heights, Queensland
  - The Skin Centre, Benowa, Queensland
  - Siller Medical, Brisbane, Queensland
- New Zealand (3):
  - Auckland Dermatology, Epsom, Auckland
  - Tristram Clinic, Hamilton
  - Skin Centre, Tauranga

REFERENCES:
- See also: Central HREC — http://www.bellberry.com.au